CLINICAL TRIAL: NCT06368128
Title: Climbing Lifestyle Intervention for Modifying Physical Activity Behaviors (CLIMB): Pilot Study
Brief Title: Climbing Lifestyle Intervention for Modifying Physical Activity Behaviors: Pilot Study
Acronym: CLIMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Michigan University (Other)
Responsible Party: Principal Investigator, Megan C. Nelson, Assistant Professor, Northern Michigan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-24_51
Record Dates: First submitted 2024-03-18; First posted 2024-04-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lifestyle Factors; Physical Inactivity; Quality of Life
Keywords: Rock Climbing; Cardiovascular Disease Risk Factors; Physical Inactivity; Quality of Life
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with participants allocated to either a control or intervention group; comparison between groups and within groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control arm will be asked to maintain their current lifestyle behaviors.
- Intervention (Experimental): Participants in the intervention arm will be asked to partake in a 12-week progressive, supervised, indoor rock climbing training program.
  Interventions: Behavioral: Indoor Rock Climbing Exercise Training Program

INTERVENTIONS:
Behavioral: Indoor Rock Climbing Exercise Training Program — Training will occur 2-3 days per week for 60 minutes; ratings of perceived exertion between 3-7 on a scale of 0-10 will be targeted for the desired intensity throughout the program. Minutes of rock climbing will also be monitored to develop the progression strategy.
  Arms: Intervention

SUMMARY:
The aim of this pilot study is to determine the effects of a 12-week indoor rock climbing training program on heart health, mental health, and behavioral health in generally healthy adults aged 18-35 years old who do not exercise. Participants will learn to rock climb using ropes on an indoor rock climbing wall and participate in the training program 2-3 days per week for 60 minutes each session over 12 weeks. Health outcomes will be measured at 4 time points over the course of the study (pre-intervention, 6-weeks/mid-intervention, 12-weeks/post-intervention, and 24-weeks post-intervention).

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of a 12-week progressive, supervised indoor rock climbing intervention on physical, mental, and behavioral health outcomes in physically inactive adults. This will be a pilot study used for informing a larger, randomized controlled trial. Measurements include: cardiometabolic disease risk factors (e.g., blood pressure, fasting glucose and lipids, hemoglobin a1c), health-related components of physical fitness (e.g., cardiorespiratory fitness, muscular fitness, dynamic balance, body composition), health-related quality of life, and behavior change variables (e.g., attitudes toward physical activity, self-efficacy for exercise, objective physical activity and sedentary behavior). The majority of rock climbing-related studies focus on enhancing performance in high-level climbing athletes and very little research has examined the specific impact of climbing physical activity on cardiovascular health parameters. Indoor climbing has demonstrated to be an activity that is safe for many individuals and does not require a high level initial fitness to partake in the activity. This study will engage generally healthy, physically inactive adults (aged 18-35 y) in an indoor rock climbing program 2 times per week for 60 minutes for the first 4 weeks and progressing to 3 times per week for 60 minutes for the last 8 weeks. Participants will partake in top-rope style rock climbing and bouldering. Data collection will occur over three visits to the School of Health and Human Performance Research Lab at four time points throughout the course of the study (baseline/pre-intervention, 6-weeks/mid-intervention, 12-weeks/post-intervention, 24-weeks post-intervention; total of 12 data collection visits).

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive
* Membership to Physical Education Instructional Facility at Northern Michigan University
* No/very little experience with rock climbing
* No diagnosed cardiovascular, metabolic, renal disease
* No current injury

Exclusion Criteria:

* Physically active
* Experience with rock climbing
* No current membership with Physical Education Instructional Facility at Northern Michigan University
* Pregnant and/or breastfeeding
* Diagnosis of cardiovascular disease, metabolic disease, renal disease
* Current or previous injury that would be exacerbated by rock climbing
* Other diagnosed conditions in which rock climbing would be contraindicated

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting lipids | 0, 6, 12, 24 weeks
  HDL-c; LDL-c; total cholesterol, triglycerides measured via capillary blood sample and point-of-care testing
Fasting glucose | 0, 6, 12, 24 weeks
  glucose (mg/dL) measured via capillary blood sample and point-of-care testing
Hemoglobin a1c | 0, 6, 12, 24 weeks
  Glycosylated hemoglobin (%) measured via capillary blood sample and point-of-care testing

SECONDARY OUTCOMES:
Physical activity and sedentary behavior | 0, 6, 12, 24 weeks
  Objectively monitored light, moderate, and vigorous physical activity minutes per week
Sedentary behavior bouts (30 min, 60 min, >60 min) | 0, 6, 12, 24 weeks
  Objectively monitored number of bouts of sedentary behavior occurring in bouts of 30 minutes or less, 30-60 minutes, and greater than 60 minutes
Cardiorespiratory fitness | 0, 12 weeks
  VO2max (mL/kg/min) measured via expired air analysis
Muscular fitness | 0, 12 weeks
  Maximal isometric handgrip strength (kg) using an electronic handgrip dynamometer
Handgrip strength asymmetry | 0, 12 weeks
  Maximal isometric handgrip strength measured using an electronic handgrip dynamometer on both hands
Lower-body dynamic balance | 0, 12 weeks
  Lower-quarter y-balance test distance (cm) on each leg, in the anterior, posteromedial, and posterolateral directions.
Health-related quality of life using CDC Health-Related Quality of Life Scale | 0, 6, 12, 24 weeks
  Core healthy days module, activity limitations module. Core healthy days module measures the number of days over the past 30 days where injury, mental health, was not good and kept individuals from performing usual activities. Activity limitations asks if individuals are limited by any health problems, how many days they are limited by health problems, and if needs are impaired. Healthy days symptom module asks if pain, depression, anxiety and sleep were an issue on any number of days over the past 30 days. Additionally, how many days individuals felt healthy and full of energy over the past 30 days.
Exercise self-efficacy measured via Self-efficacy for exercise scale | 0, 6, 12, 24 weeks
  Self-efficacy for exercise scale is 9 items representing various scenarios that are measured on a scale of 1 (not confident) to 10 (very confident) a participant feels to exercise in that scenario. Higher scores represent higher self-efficacy for exercise participation.
Perceptions of exercise measured via Views and Attitudes Toward Exercise Scale | 0, 6, 12, 24 weeks
  Views and attitudes towards exercise scale is 15 items measured on a 7-point Likert scale from strongly disagree (lowest) to strongly agree (highest). Sum up all responses, higher scores are better perceptions of exercise.
Perceived stress | 0, 6, 12, 24 weeks
  Perceived stress scale items are scored from adding up each alternative over 10 items: 0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often. 0-13=low stress, 14-26=moderate stress, 27-40=high perceived stress.
Blood pressure | 0, 6, 12, 24 weeks
  Systolic and diastolic blood pressure (mmHg) measured via automated blood pressure cuff.
Body composition | 0, 12, 24 weeks
  Fat free mass, fat mass in kg using Dual-energy x-ray absorptiometry
Bone density | 0, 12, 24 weeks
  Total bone density (g/cm3) using Dual-energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Megan C Nelson, PhD, Principal Investigator — Northern Michigan University
Locations (1):
- Northern Michigan University, Marquette, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study; individual participant data will not be shared to protect participants information so that it remains confidential.